CLINICAL TRIAL: NCT05218707
Title: Influence of Oropharyngeal Airway on the Incidence of Airway Complications Following LMA Removal Under Deep Anaesthesia in Children
Brief Title: Oropharyngeal Airway and Airway Complications
Status: Recruiting | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Khalid Siddiqui, Assistant Professor, Aga Khan University
Other Study IDs: 2021-5669-19713
Record Dates: First submitted 2022-01-31; First posted 2022-02-01 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Airway Complication of Anesthesia
Keywords: laryngeal mask airway; Oropharyngeal Airway; Deep Anaesthesia; Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: An appropriate size oropharyngeal airway (GUEDEL) will be inserted immediately after removal of LMA and time will be noted. (Size will be chosen by placing the flange at the corner of the mouth and tip at the angle of the jaw).
  Interventions: Other: GUEDEL Airway
- Group B: In Group B No oropharyngeal airway (GUEDEL) will be inserted.

INTERVENTIONS:
Other: GUEDEL Airway — GUEDEL Airway of size '000,00,0,' and '1' will be used.
  Groups: Group A

SUMMARY:
Laryngeal Mask Airway has been used in paediatric anaesthesia since the 1990's. Clinical practice in paedeatric anaesthesia for Laryngeal Mask Airway removal varies and there is no standard of care.

In children removing the Laryngeal Mask Airway under deep inhalational anaesthesia has some advantages compared to awake, but may be associated with higher rate of complications when Laryngeal Mask Airway is removed in supine compared to lateral position. On the other hand deep anaesthesia may cause airway obstruction due to reduction in tone of upper airway muscles in some patients. An oropharangeal airway may prevent this. This aspect had not been studied before and represent a gap in literature.

Study Hypothesis:

Airway complications associated with Laryngeal Mask Airway removal under deep anaesthesia are same with or without insertion of an oral airway. Alternate hypothesis is that airway complications be less if an air way is inserted at the end of anaesthesia.

Objective:

The present study was designed to observe any difference in immediate complication after removal of LMA in supine head down position under deep anaesthesia with or without insertion of an oro-pharyngeal airway. Airway complications that we will observe are desaturation <92%, stridor, excessive secretions, laryngospasm, retching, vomiting, coughing, trauma to the soft tissues and damage to the teeth.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients aged 2-10 years undergoing surgery where anaesthesia with LMA is considered appropriate.

Exclusion Criteria:

* Patients undergoing surgery involving soiling of the airway
* Patients with conditions associated with higher incidence of gastrooseophageal reflux
* Presence of active upper respiratory tract infection (URI)
* Emergency Surgery

Ages: 2 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Children aged 2-10 years undergoing surgery where anaesthesia with Laryngeal Mask Airway insertion.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation | Day 1
  Oxygen saturation <92% will be considered as complication
Stridor | Day 1
  The presence of noisy breathing occurring through obstructed airflow. We clinically measure it by auscultation of the nose, oropharynx, neck and chest.

SECONDARY OUTCOMES:
laryngospasm | Day 1
  The occurrence of a transient and reversible spasm of the vocal cords. We will evaluate laryngospasm by observing a high pitch inspiratory stridor followed by partial or complete airway obstruction.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mason DG, Bingham RM. The laryngeal mask airway in children. Anaesthesia. 1990 Sep;45(9):760-3. doi: 10.1111/j.1365-2044.1990.tb14449.x. PMID 2100990
- [Background] Thomas-Kattappurathu G, Kasisomayajula A, Short J. Best position and depth of anaesthesia for laryngeal mask airway removal in children: A randomised controlled trial. Eur J Anaesthesiol. 2015 Sep;32(9):624-30. doi: 10.1097/EJA.0000000000000286. PMID 26086281
- [Background] Sinha A, Sood J. Safe removal of LMA in children - at what BIS? Paediatr Anaesth. 2006 Nov;16(11):1144-7. doi: 10.1111/j.1460-9592.2006.01978.x. PMID 17040303